CLINICAL TRIAL: NCT06931730
Title: Reprogramming Energy Homeostasis in Overweight Children and Adults Trough Exercise, Cognitive Training and Social Interaction
Brief Title: Reprogramming Energy Homeostasis in Overweight Individuals Via Exercise, Cognitive, and Social Training
Acronym: Resilient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Melania Manco, Medical Director, Preventive and Predictive Medicine, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-MAD-2022-12376459
Record Dates: First submitted 2025-03-24; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Overweight; Leptin Resistance; Childhood Obesity
Keywords: childhood obesity; cognitive training; social training; environmental enrichment; leptin; lifestyle modification; overweight; obesity; energy expenditure; thermogenesis; physical activity; leptin sensitivity; leptin resistance
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intensive Health Behavior Treatment group: Physical Activity and Diet (Active Comparator): Participants will be provided with a personalized dietary plan and a Physical Activity training
  Interventions: Other: Nutritional Intervention; Other: Physical Activity training
- Cognitive Training group: Physical Activity, Diet and an online cognitive training (Active Comparator): Participants will be provided with personalized dietary plan, a Physical Activity training, and an online cognitive training.
  Interventions: Other: Nutritional Intervention; Other: Physical Activity training; Other: Cognitive training
- Social Training group: Physical Activity, Diet and cognitive training (Active Comparator): Participants will be provided with personalized dietary plan, a Physical Activity training, and a peer interaction program in ecological context.
  Interventions: Other: Nutritional Intervention; Other: Physical Activity training; Other: Social Training

INTERVENTIONS:
Other: Nutritional Intervention — Participants will receive comprehensive dietary education from the nutritionists of the research team, aimed at improving their baseline diet by incorporating nutritional recommendations based on the Mediterranean diet and the Italian dietary guidelines for healthy eating.
Other: Physical Activity training — Participants will engage in a structured exercise program designed to improve motor competence and confidence. Tailored to each individual's baseline physical abilities and cardiorespiratory capacity, the program will focus on enhancing aerobic fitness, flexibility, and coordination.
Other: Cognitive training — Participants will undergo an online cognitive training program, with a particular focus on memory enhancement.
  Arms: Cognitive Training group: Physical Activity, Diet and an online cognitive training
Other: Social Training — A peer interaction program within an ecological setting, meant as a natural context of daily life, will be offered to participants. The program aims to improve active listening skills, comprehension of various communication styles (passive, assertive, aggressive), and the efficient recognition and management of emotions.
  Arms: Social Training group: Physical Activity, Diet and cognitive training

SUMMARY:
The RESILIENT project is a clinical trial investigating leptin sensitivity in both children and adults with overweight or obesity. The study examines the additive effects of Cognitive Training (CT) and Social Training (ST) on leptin sensitivity, compared to stand-alone Intensive Health Behaviour Treatment (IHBT), which includes diet and Physical Activity (PA).

The intervention will last for 8 weeks, followed by a 12-week washout period. A multilevel assessment will be conducted, evaluating in vivo leptin sensitivity (through the ratio of leptin levels to caloric intake) as well as ex vivo molecular analysis of leptin signaling in Peripheral Blood Mononuclear Cells (PBMCs). Additionally, clinical, psychological, cognitive, and physiological assessments will be performed to assess the efficacy of each intervention. By investigating leptin resistance as a potential molecular bridge between metabolic dysregulation and cognitive dysfunctions, this study may contribute to the development of more effective, long-term treatments for obesity and overweight. Additionally, in vivo investigation of leptin sensitivity may be particularly important for providing evidence of the metabolic and cognitive effects necessary for developing novel anti-obesity treatments.

ELIGIBILITY:
Inclusion Criteria:

* a condition of overweight or obesity
* Intelligence Quotient (IQ) ≥ 85

Exclusion Criteria:

* genetic or syndromic obesity;
* reduced mobility;
* systemic diseases;
* ongoing pharmacological treatment for chronic conditions.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
In Vivo Leptin Sensitivity | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Leptin sensitivity will be evaluated as the ratio between caloric intake during an experimental meal and circulating leptin levels. Participants will receive a standardized breakfast and after 3 hours an ad libitum lunch, with detailed records of consumption, additional food requests, and portion sizes. Hunger and satiety will be measured using a 5-item Visual Analogue Scale (VAS) at multiple time points, recorded in millimeters. Energy and nutrient intake will be assessed using nutritional labels from each food item, and leptin sensitivity will be determined via plasma fasting.
Ex Vivo Leptin Sensitivity | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Since direct assessment of leptin sensitivity in the central nervous system is not feasible in humans, peripheral leptin sensitivity ex vivo will be evaluated using Peripheral Blood Mononuclear Cells (PBMCs). PBMCs will be collected from the same individuals before and after the intervention and exposed to recombinant leptin to assess intracellular signalling activation. The primary leptin effector pathway is Janus kinase 2/signal transducer and activator of transcription 3 (JAK2/STAT3), though Extracellular signal-regulated protein kinases 1 and 2 (ERK1/2) activation has also been reported among others. The activation of these pathways will be measured using immunoassays such as Enzyme Linked Immunosorbent Assay (ELISA) and Western blot, quantifying the ratio of phosphorylated to total protein levels for each intracellular effector.
Insulin Sensitivity and Secretion | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Insulin sensitivity and secretion will be assessed both during fasting and the oral glucose tolerance test (OGTT).
Energy Metabolism | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Energy metabolism, including resting metabolic rate and diet-induced thermogenesis, will be measured by indirect calorimetry.
Fat Mass (percentage) | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Fat mass will be estimated using bioelectrical impedance analysis and expressed as a percentage of total body weight.
Fat Mass (kilograms) | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Fat mass will be estimated using bioelectrical impedance analysis and expressed in kilograms.

SECONDARY OUTCOMES:
Non-Verbal Fluid Intelligence | At baseline (T0)
  Assessed using the Colored Progressive Matrices (CPM), a standardized test that measures the ability to recognize patterns and solve problems without reliance on language. The outcome is the global Intelligent Quotient (IQ) score, with a mean of 100 and a standard deviation of 15, measured in standardized scores.
Working Memory | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Evaluated through the N-Back Task, a computerized assessment of both visuo-spatial and verbal working memory. In the visuo-spatial condition, participants view randomly positioned blue boxes and determine whether the current position matches the previous one. In the verbal condition, they listen to a stream of letters and identify whether each letter matches the one immediately preceding it. The task adapts dynamically, increasing in difficulty when accuracy reaches or exceeds 80%. The outcome metric is the accuracy percentage at each difficulty level, measured in percentage of correct responses.
Sustained Attention and inhibitory control | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Measured using the Continuous Performance Test-II (CPT-II), a computerized assessment of sustained attention and inhibitory control. Participants respond to any letter except "X" (Go trials) and withhold responses when "X" appears (No-Go trials). Reaction times and response variability provide insights into attentional performance. The outcome metrics include accuracy, reaction time (RT) in milliseconds, and reaction time variability (RTV) in milliseconds.
Episodic Long-Term Memory | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  To assess episodic long-term memory, the Verbal and Visual-Spatial Learning tasks from the standardized Battery for the evaluation of Memory (PROMEA) will be administered. The Verbal Learning Task presents a list of 15 unrelated words across 3 trials, followed by delayed recall after 15 minutes. Similarly, the Visual-Spatial Learning Task involves recalling the placement of 15 objects in 4 quadrants during 3 trials, with delayed recall after 15 minutes. The outcome metrics include the number of words or objects recalled across trials and the delayed recall score, expressed in standard scores and percentile ranks.
Visual-Motor Integration | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Assessed using the Test of Visual Motor Integration (VMI), which evaluates the coordination between visual perception and motor function. It consists of 3 components: Visual Motor Integration, requiring participants to copy increasingly complex forms; Visual Perception, involving the identification of matching forms among distractors; and Fine Motor Coordination, assessing precision in connecting dots within defined boundaries. The outcome includes raw scores converted to standard scores, with a mean of 100 and a standard deviation of 15, as well as percentile ranks.
Gross and Fine Motor Skills | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Measured using the Movement Assessment Battery for Children-2 (MABC-2), which evaluates motor skills through 3 components: Manual Dexterity, assessing fine motor control; Aiming and Catching, measuring coordination between fine and gross motor movements; and Balance, which examines static and dynamic postural control through structured physical tasks. The outcomes are expressed as standard scores (mean = 100, SD = 15) and percentile ranks.
Short-Term Memory | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Evaluated using the Battery for Neuropsychological Evaluation of Children Battery (BVN 5-11), including the Digit Span and Corsi Block-Tapping Tests. The Digit Span Test requires participants to repeat sequences of numbers in the same or reversed order, assessing verbal short-term memory. The Corsi Block-Tapping Test involves replicating sequences of tapped blocks to assess visuo-spatial short-term memory. The score is determined by the number of items correctly recalled, expressed as Z-scores based on a normative sample, where a Z-score of 0 indicates the average performance of the normative group.
Behavioral and Emotional Symptoms | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Assessed using the Child Behavior Checklist for Ages 6-18 (CBCL 6-18), a standardized parent-report questionnaire, comprised of 8 syndrome scales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behaviour, and aggressive behaviour), 3 broadband scores (internalizing and externalizing problems, and total problem), Diagnostic and Statistical Manual of mental disorders (DSM)-oriented scales (affective problems, anxiety problems, somatic problems, attention deficit/hyperactivity problem, oppositional defiant problems, conduct problems), and the 2007 Scales (sluggish cognitive tempo, obsessive-compulsive problems, post-traumatic stress problems). For each subscale raw scores will be converted in T-scores (M = 50, SD = 10).
Ankle Dorsiflexion | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Ankle dorsiflexion will be evaluated using the Knee to Wall test, in which the participant places one foot touching the wall and gradually moves back until being able to touch the wall with the knee while keeping the heel on the ground.
Joint Mobility | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Joint mobility will be assessed through a Scapular-Humeral Circumduction test, conducted with a calibrated stick, where the result is the last completed circumduction with extended arms.
Trunk Strength | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Trunk strength will be assessed using the Trunk Lift test, in which participants lie prone on a mat and lift their upper body off the floor to their maximum height. The distance between the floor and the participant's chin will be measured.
Flexibility: Sit and Reach Test | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  In the Sit and Reach test, participants sit with their legs extended and feet dorsiflexed against a 30 cm support, then perform a forward trunk flexion. The result is measured as the distance between the fingertips and the toes.
Flexibility: Lateral Trunk Flexion Test | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Flexibility will also be assessed using the Lateral Trunk Flexion test, which records the difference between the initial hand position and the maximum lateral flexion.
Quality of Life: Physical, Emotional, Social, and School Functioning | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  The Pediatric Quality of Life Inventory (PedsQL version 4) is a widely used tool in studies involving children with obesity to measure key dimensions of health and quality of life. It includes domains of Physical, Emotional, Social, and School Functioning. Both child self-report and parent-report formats will be administered. Total Score and Psychosocial Health Summary Score will be calculated as percentages. Higher percentages indicate better functioning across these domains.
Social Adaptive Skills | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  The social skill domain will be investigated through the standardized parent-reported Adaptive Behavior Assessment System, Second Edition (ABAS-II), which will provide the Social Adaptive Composite (SAC), which summarizes performance across the Leisure and Social skill areas. Raw scores will be converted into standardized weighted scores (M = 10, SD = 3) and standard scores (M = 100, SD = 15).
Social Skills | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  The Social Responsiveness Scale (SRS) will be used as well. The SRS is a standardized parent-report measure frequently used with children and adolescents between the ages of 4 and 18 years to screen subtle social communication deficits. The SRS generates 5 subscales: social awareness, social cognition, social motivation and social communication. Raw scores will be converted to gender-normed T-scores (M = 50, SD = 10).
Eating Behavior and Disorders | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  The Eating Disorders Questionnaire in Childhood (EDQ-C) is a standardized tool used for the early identification of eating disorders in children, assessing comorbidities with attachment patterns, anxiety and mood disorders, as well as relational and behavioural difficulties. It includes a self-report version for children aged 8 and older, and 2 parent-report forms based on the child's age (4-7 and 8-12 years). For each diagnostic category, raw scores will be calculated and converted into standard score and percentile ranks (< 90 = within normal range, > 95 = clinically significant, > 99 = pathological).
Sleep Habits and Quality | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  To assess sleep habits and quality, the Sleep Disturbance Scale for Children (SDSC) will be employed. This standardized parent-report questionnaire evaluates various aspects of children's sleep, including duration, onset time, sleep disorders and an overall measure of sleep disturbances in children and adolescents aged 6 to 15 years. Six main areas are investigated by the following subscales: Disorders in Initiating and Maintaining Sleep (DIMS), Sleep Breathing Disorders (SBD), Arousal Disorders (DA), Sleep-Wake Transition Disorders (SWTD), Excessive Sleepiness (DES), and Nocturnal Hyperhidrosis (NH). For each subscale raw scores will be converted in T-scores (M = 50, SD = 10).
Brain Function | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Brain responses will be studied through vascular brain activity to a glucose challenge, measured using functional near-infrared spectroscopy (fNIRS) in children and functional MRI (fMRI) in adults.
Plasma Analysis | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Plasma samples will be analysed for circulating levels of adipokines and cytokines (R&D Systems, Inc. 614 McKinley Place NE Minneapolis, MN 55413), including Brain-Derived Neurotrophic Factor (BDNF), a key regulator of neural plasticity and appetite suppression, Pro-OpioMelanoCortin (POMC) and its derivative Melanocyte-Stimulating Hormone (MSH), which play a central role in the anorectic response to leptin, eotaxin/CCL11, a proinflammatory chemokine linked to age-related cognitive decline, and Insulin-like Growth Factor-Binding Protein 2 (IGFBP2), a liver-derived protein regulated by leptin and involved in glucose homeostasis.
Gut Microbioma | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  The composition of the gut microbiota will be assessed using genomic analysis of stool samples collected from participants. Fresh stool samples will be collected by participants at home, immediately frozen at approximately -20°C, and transported in a refrigerated box to the biobank. Upon arrival, the samples will be stored at -80°C until DNA extraction.
Muscle Strength: Upper Limb Strength | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Upper limb strength will be evaluated with a Floor Press test using calibrated dumbbells based on each participant's strength.
Muscle Strength: Handgrip Strength | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Handgrip strength will be assessed using a dynamometer.
Lower Limb Explosive Strength | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Lower limb explosive strength will be measured with the Standing Long Jump test, where participants jump as far as possible, landing with both feet together; the best of two attempts will be considered.
Abdominal Strength and Endurance | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Abdominal strength and endurance will be assessed with a Sit-Up test, where participants lie supine with their legs bent at 90° and perform sit-ups, with the result being the maximum number of repetitions performed.
Balance | At baseline (T0), at the end of the 8-week intervention (T1, end of month 2), and 12 weeks after the intervention (T2, end of month 5) to verify the persistence of effects.
  Balance will be assessed using the Single Leg Stance test, where participants maintain a single-leg stance within a shoe-sized rectangle for 60 seconds, with the number of falls recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Rome, Italy
  - Bambino Gesù Hospital and Research Institute,, Rome, Rome

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request, subject to validation by the OPBG Ethics Committee, in compliance with GDPR and European regulations. Alternatively, aggregated data may be considered.
Supporting Information: Study Protocol
Time Frame: The time frame for data availability will be determined in accordance with GDPR and relevant European regulations.
Access Criteria: Access to the IPD and supporting information will be granted to the Principal Investigator (PI) of the research, Dr. Melania Manco (melania.manco@opbg.net).
URL: https://www.ospedalebambinogesu.it/ospedale/comitato-etico/

REFERENCES:
- [Derived] Russo V, Menghini D, Mainardi M, Fintini D, Aureli A, Gianni N, Rava L, Rea MA, Scozia G, Spiezia C, Scabia G, Furini G, Vicari S, Cianfarani S, Maffei M, Manco M. Reprogramming energy homeostasis in children with overweight through cognitive training and social interaction. A study protocol to estimate leptin sensitivity. Front Endocrinol (Lausanne). 2025 Jun 18;16:1606132. doi: 10.3389/fendo.2025.1606132. eCollection 2025. PMID 40607230